CLINICAL TRIAL: NCT06130020
Title: Comparing Targets of Expressive Writing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Princeton University (Other)
Responsible Party: Principal Investigator, Erik Nook, Assistant Professor, Trustees of Princeton University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Princeton15734
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Anxiety; Depression
Keywords: expressive writing; journaling; mental health
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Self (Experimental): The Self group is instructed to carry out the expressive writing exercise as if they were writing to themselves.
  Interventions: Behavioral: Expressive Writing: Self
- Other (Experimental): The Other group is instructed to carry out the expressive writing exercise as if they were writing to someone they feel close to.
  Interventions: Behavioral: Expressive Writing: Other
- Control (Placebo Comparator): The Control group is asked to write down a factual description of their routine that day, as if they were writing to themselves.
  Interventions: Behavioral: Factual Writing

INTERVENTIONS:
Behavioral: Expressive Writing: Self — This intervention consists of a daily expressive writing exercise carried out for 14 consecutive days, for 15 minutes each day. Expressive writing involves asking participants to write about their deepest thoughts and feelings surrounding an emotional event. Participants in this condition will write as if they are writing to themselves.
  Arms: Self
Behavioral: Expressive Writing: Other — This intervention consists of a daily expressive writing exercise carried out for 14 consecutive days, for 15 minutes each day. Expressive writing involves asking participants to write about their deepest thoughts and feelings surrounding an emotional event. Participants in this condition will write as if they are writing/talking to someone they're close to.
  Arms: Other
Behavioral: Factual Writing — This intervention consists of a daily factual writing exercise carried out for 14 consecutive days, for 15 minutes each day. Participants are asked to give a factual description of their day. This is a standard control for Expressive writing studies. Participants in this condition will be asked to direct their writing to themselves.
  Arms: Control

SUMMARY:
Expressive writing involves writing about one's deepest thoughts and feelings surrounding an emotional event. The current literature on the efficacy of expressive writing is mixed and warrants further investigation into how, when, and for whom expressive writing is an effective intervention. The goal of this study is to compare the efficacy of expressive writing interventions in young adults when people imagine that they're writing to themselves vs. a loved one. Participants will carry out an expressive writing exercise for 14 consecutive days. Participants are randomized into 3 groups: Self, Other, and Control. The Self group is instructed to write as if they were talking to themselves. The Other group is instructed to direct their writing to someone they feel close to. The Control group is asked to write down a factual description of their routine that day, and direct this writing to themselves. We will recruit participants until we have usable data from 53 participants per group (i.e., 159 in total).

ELIGIBILITY:
Inclusion Criteria:

* US-based
* Fluent English
* Combined GAD-7 and PHQ-8 score of ≥ 5

Exclusion Criteria:

* "Completion" of a writing session requires participants to spend at least 15 minutes on the writing page. We will monitor completion of the daily writing exercise, and will contact participants who miss or spend less than 15 minutes on the exercise. Participants who fail to complete 3 consecutive daily writing sessions will be deemed non-compliant, removed from the study, and paid a prorated amount for the tasks they have completed in the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Initial visit (day 1), mid-point (day 7) final visit (day 15), 1-month follow-up (1 month after day 14)
  Generalized Anxiety Disorder-7 (GAD-7). Scores range from 0-21, with higher scores indicating more severe anxiety.
Depression | Initial visit (day 1), mid-point (day 7), final visit (day 15), 1-month follow-up (1 month after day 14)
  Patient Health Questionnaire-8 (PHQ-8). Scores range from 0-24, with higher scores indicating more severe depression.

OTHER OUTCOMES:
Sleep Quality | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Pittsburgh Sleep Quality Index (PSQI). Total scores range from 0-21, with higher scores indicating poorer sleep quality.
Depression, Anxiety, and Stress | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Depression, Anxiety, and Stress-21 (DASS-21). Scores for each of the three subscales range from 0-42, with higher scores indicating greater severity.
Alexithymia (TAS) | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Toronto Alexithymia Scale-20 (TAS-20). Scores range from 20-100, with higher scores indicating greater alexithymia.
Alexithymia (PAQ) | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Perth Alexithymia Questionnaire (PAQ). Total scores range from 24-168, with higher scores indicating greater alexithymia.
Emotion Regulation | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Emotion Regulation Questionnaire (ERQ). Scores for the reappraisal and suppression subscales range from 6-42 and 4-28 respectively. Higher scores indicate greater use of the strategy.
Interpersonal Regulation | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Interpersonal Regulation Questionnaire (IRQ). Total scores range from 16-112, with higher scores indicating greater tendency to use/efficacy of interpersonal emotion regulation.
Social Desirability | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Marlow-Crowne Social Desirability Scale (MC-SDS). Scores range from 0-33, with higher scores indicating greater social desirability.
Social Connectedness | Initial visit (day 1), final visit (day 15), 1-month follow-up (1 month after day 14)
  Social Connectedness Scale (SCS). Scores range from 8-48, with higher scores indicating greater connectedness to others.
Daily Sleep | Daily from day 1 to day 14
  Consensus Sleep Diary (CSD). Items are used to derive estimates of sleep indices, such as time in bed and total sleep time.
Sleepiness | Daily from day 1 to day 14
  Karolinska Sleepiness Scale (KSS). Scores on this single-item scale range from 1-10, with higher scores indicating greater sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Nook, PhD, Principal Investigator — Princeton University
Locations (1):
- Peretsman Scully Hall, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion, a subset of the de-identified data will be transferred to OSF, which will provide public access to this data. Writing content will not be transferred to OSF, though we will make thoroughly de-identified data available to researchers who have completed appropriate ethics training, agree to confidentiality restrictions, and whose research goals are in line with the purpose of this study.
Supporting Information: SAP, Analytic Code
Time Frame: Beginning after publication of results with no end date.
Access Criteria: A subset of the de-identified data will be publicly available on the OSF.

REFERENCES:
- [Background] Pennebaker JW, Beall SK. Confronting a traumatic event: toward an understanding of inhibition and disease. J Abnorm Psychol. 1986 Aug;95(3):274-81. doi: 10.1037//0021-843x.95.3.274. No abstract available. PMID 3745650